CLINICAL TRIAL: NCT00546364
Title: IXTEND: A Randomized Phase 2 Study to Evaluate the Combination of Ixabepilone Plus Capecitabine or Capecitabine Plus Docetaxel in the Treatment of Metastatic Breast Cancer
Brief Title: Randomized Study Evaluating Ixabepilone Plus Capecitabine or Docetaxel Plus Capecitabine in Metastatic Breast Cancer
Acronym: IXTEND
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: R-Pharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA163-131
Record Dates: First submitted 2007-10-17; First posted 2007-10-18 (Estimated); Results first posted 2011-06-01 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-02

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — ixabepilone; Capecitabine; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ixabepilone, 40 mg/m^2 + Capecitabine, 1000 mg/m^2 (Experimental)
  Interventions: Drug: Ixabepilone, 40 mg/m^2 + Capecitabine, 1000 mg/m^2
- Ixabepilone, 32 mg/m^2 + Capecitabine, 1000 mg/m^2 (Experimental)
  Interventions: Drug: Ixabepilone, 32 mg/m^2 + Capecitabine, 1000 mg/m^2
- Docetaxel, 75 mg/m^2 + Capecitabine, 1000 mg/m^2 (Active Comparator)
  Interventions: Drug: Docetaxel, 75 mg/m^2 + Capecitabine, 1000 mg/m^2

INTERVENTIONS:
Drug: Ixabepilone, 40 mg/m^2 + Capecitabine, 1000 mg/m^2 — Ixabepilone, 40 mg/m^2, administered as a 3-hour intravenous (IV) infusion on Day 1 of a 21-day cycle plus capecitabine, 1000 mg/m^2, self-administered on an outpatient basis twice daily by mouth on Days 1 through 14 (±2 days) of each 21-day cycle.
  Other Names: IXEMPRA®; BMS-247550
  Arms: Ixabepilone, 40 mg/m^2 + Capecitabine, 1000 mg/m^2
Drug: Ixabepilone, 32 mg/m^2 + Capecitabine, 1000 mg/m^2 — Ixabepilone, 32 mg/m^2, administered as a 3-hour IV infusion on Day 1 of a 21-day cycle plus capecitabine, 1000 mg/m^2, self-administered on an outpatient basis twice daily by mouth on Days 1 through 14 (±2 days) of each 21-day cycle.
  Arms: Ixabepilone, 32 mg/m^2 + Capecitabine, 1000 mg/m^2
Drug: Docetaxel, 75 mg/m^2 + Capecitabine, 1000 mg/m^2 — Docetaxel 75 mg/m^2 administered as a 1-hour IV infusion on Day 1 of a 21-day cycle plus capecitabine, 1000 mg/m^2, self-administered on an outpatient basis twice daily by mouth on Days 1 through 14 (±2 days) of each 21-day cycle.
  Arms: Docetaxel, 75 mg/m^2 + Capecitabine, 1000 mg/m^2

SUMMARY:
The purpose of this study is to assess the effect of ixabepilone plus capecitabine or docetaxel plus capecitabine on shrinking or slowing the growth of metastatic breast cancer in women. The safety of this combination therapy will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Participants with metastatic breast cancer
* Measurable disease
* Up to 1 chemotherapy regimen is acceptable. Participants who have received paclitaxel in the neoadjuvant or adjuvant setting acceptable, only if the last dose of paclitaxel was received 12 months or less before the treatment. There is no timeframe for prior paclitaxel in the metastatic setting.
* Human epidermal growth factor receptor 2-positive participants allowed if they have progressed after receiving treatment with trastuzumab or lapatinib
* Eastern Cooperative Oncology Group Performance status of 0-1
* Age younger than 18 years
* Women of childbearing potential must be using an adequate method of contraception to avoid pregnancy throughout the study and for at least 4 weeks after the last dose of investigational products

Exclusion Criteria:

* More than 1 chemotherapy regimen for the treatment of metastatic breast cancer
* Prior treatment with any epothilone, capecitabine, or docetaxel
* Prior radiation must not have included 30% or more of major bone marrow-containing areas (pelvis, lumbar spine). If prior radiation was less than 30%, a minimum interval of 2 weeks must be allowed between the last radiation treatment and administration of study medication. There must be at least 1 week between focal/palliative radiation and administration of study medication.
* Any current or previous history of brain and/or leptomeningeal metastases
* Neuropathy greater than Grade 2
* Any concurrent malignancy other than nonmelanoma skin cancer or carcinoma in situ of the cervix
* Uncontrolled diabetes mellitus
* Chronic hepatitis
* HIV-positive status
* Administration of trastuzumab, lapatinib, bevacizumab, or other systemic treatment for cancer must be discontinued 28 days prior to study medication. Hormonal anticancer agents must be discontinued at least 14 days prior to study medication. Hormonal replacement therapy is acceptable
* Biphosphonates for palliation of bone metastases allowed if initiated at least 7 days before study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2008-02; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (60):
- United States (60):
  - Dch Cancer Treatment Center, Tuscaloosa, Alabama
  - Scripps Cancer Center, La Jolla, California
  - Cancer Center of Central Connecticut, Southington, Connecticut
  - Local Institution, Newark, Delaware
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Local Institution, Jacksonville, Florida
  - Local Institution, Miami, Florida
  - Medical Oncology Associates of Augusta, PC, Augusta, Georgia
  - Local Institution, Honolulu, Hawaii
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - John W Kugler, MD, Peoria, Illinois
  - Midwestern Regional Medical Center, Zion, Illinois
  - Center for Cancer Care at Goshen Health System, Goshen, Indiana
  - Monroe Medical Associates, Munster, Indiana
  - Cancer Center of Kansas, Wichita, Kansas
  - University of Kentucky, Lexington, Kentucky
  - University Medical Center, Inc, Louisville, Kentucky
  - Hematology/Oncology Clinic, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Center for Cancer & Blood Disorders, PC, Bethesda, Maryland
  - Jackson Oncology Associates, Pllc, Jackson, Mississippi
  - The Center for Cancer and Hematologic Disease, Cherry Hill, New Jersey
  - The Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Howell Office Plaza, Howell Township, New Jersey
  - Local Institution, Newark, New Jersey
  - Cooper Hospital, Division of Hematology/Oncology, Voorhees Township, New Jersey
  - UNM Cancer Center, Albuquerque, New Mexico
  - New Mexico Cancer Care Associates (NMCCA), Santa Fe, New Mexico
  - Arena Oncology Associates, PC, Lake Success, New York
  - Hematology Oncology Associates of Rockland, Nyack, New York
  - Gaston Hematology and Oncology, Gastonia, North Carolina
  - Marion L Shepard Cancer Center, Washington, North Carolina
  - Akron General Medical Center, Akron, Ohio
  - Summa Health System, Akron, Ohio
  - Local Institution, Canton, Ohio
  - Mid Ohio Oncology/Hematology, Inc, dba The Mark H Zangmeister Center, Columbus, Ohio
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Hematology & Oncology Associates of Nepa, Dunmore, Pennsylvania
  - Regional Hematology Oncology, PC, Langhorne, Pennsylvania
  - St Mary Medical Center, Langhorne, Pennsylvania
  - Local Institution, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - Local Institution, Woonsocket, Rhode Island
  - Charleston Cancer Center, Charleston, South Carolina
  - Lowcountry Hematology & Oncology, PA, Mt. Pleasant, South Carolina
  - Santee Hematology/Oncology, Sumter, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Kingsport Hematology Oncology, Kingsport, Tennessee
  - The University of Tennessee Medical Center, Knoxville, Tennessee
  - Austin Cancer Centers, Austin, Texas
  - Cancer Specialists of South Texas, Corpus Christi, Texas
  - Coastal Bend Cancer Center, Corpus Christi, Texas
  - Edward L Middleman, MD, Duncanville, Texas
  - Section Chief Medical Oncology, Houston, Texas
  - Jose A Figueroa, MD, Lubbock, Texas
  - Southlake Oncology, Southlake, Texas
  - Peninsula Cancer Institute, Newport News, Virginia
  - Providence Cancer Center, Spokane, Washington
  - Leah L Dietrich, MD, La Crosse, Wisconsin

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 62 participants enrolled, 62 were randomized and received treatment. Investigators had to terminate the study because an adequate number of participants could not be enrolled.
Groups:
- Ixabepilone, 40 mg/m^2 + Capecitabine, 1000 mg/m^2: Ixabepilone, 40 mg/m^2, administered as a 3-hour intravenous (IV) continuous infusion on Day 1 of a 21-day cycle plus capecitabine, 1000 mg/m^2, given twice daily by mouth on Days 1 through 14 (±2 days) of each 21-day cycle, self-administered on an outpatient basis.
- Ixabepilone, 32 mg/m^2 + Capecitabine, 1000 mg/m^2: Ixabepilone, 32 mg/m^2, administered as a 3-hour IV continuous infusion on Day 1 of a 21-day cycle plus capecitabine, 1000 mg/m^2, given twice daily by mouth on Days 1 through 14 (±2 days) of each 21-day cycle, self-administered on an outpatient basis.
- Docetaxel, 75 mg/m^2 + Capecitabine, 1000 mg/m^2: Docetaxel, 75 mg/m^2, administered as a 1-hour IV infusion on Day 1 of a 21-day cycle plus capecitabine, 1000 mg/m^2, given twice daily by mouth on Days 1 through 14 (±2 days) of each 21-day cycle, self-administered on an outpatient basis.
Period: Overall Study
Arm/Group | Ixabepilone, 40 mg/m^2 + Capecitabine, 1000 mg/m^2 | Ixabepilone, 32 mg/m^2 + Capecitabine, 1000 mg/m^2 | Docetaxel, 75 mg/m^2 + Capecitabine, 1000 mg/m^2
Started | 20 | 22 | 20
Never Treated | 0 | 0 | 0
Completed | 3 (Still on treatment) | 4 (Still on treatment) | 3 (Still on treatment)
Not Completed | 17 | 18 | 17
Not completed — Disease progression | 5 | 11 | 8
Not completed — Completed and off treatment | 1 | 0 | 2
Not completed — Administrative reason by sponsor | 1 | 0 | 0
Not completed — Poor compliance/noncompliance | 0 | 0 | 1
Not completed — No longer meets study criteria | 1 | 1 | 0
Not completed — Withdrawal by Subject | 5 | 6 | 3
Not completed — Prior taxotere | 1 | 0 | 0
Not completed — Mixed response | 1 | 0 | 0
Not completed — Palliative treatment | 1 | 0 | 1
Not completed — Target lesions resected | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Sponsor decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ixabepilone, 40 mg/m^2 + Capecitabine, 1000 mg/m^2 | Ixabepilone, 32 mg/m^2 + Capecitabine, 1000 mg/m^2 | Docetaxel, 75 mg/m^2 + Capecitabine, 1000 mg/m^2 | Total
Number analyzed (Participants) | 20 | 22 | 20 | 62
Age, Continuous [Median (Full Range); unit: years] | 55.5 [32 to 68] | 59 [39 to 79] | 55.5 [33 to 65] | 57.5 [32 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 22 | 20 | 62
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 4 | 4 | 13
  White | 15 | 18 | 16 | 49
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Best Tumor Response as Assessed With Response Evaluation Criteria in Solid Tumors (RECIST)
Description: RECIST definitions: Complete reponse (CR)=disappearance of all nontarget lesions; partial response (PR)=at least 30% reduction in the sum of the longest diameter (LD) of all target lesions in reference to the baseline sum LD; stable disease (SD)=neither PR nor progressive disease (PD) criteria were met; PD=at least 20% increase in the sum of the LD of all target lesions, taking as reference the smallest sum LD recorded at or following baseline. Tumor status assessed by investigator.
Time Frame: Baseline to 6 weeks (end of Cycle 2)
Population: All participants with measurable disease who have a correct cancer diagnosis and have received any treatment.
Measure: Number; unit: Participants
Arm/Group | Ixabepilone, 40 mg/m^2 + Capecitabine, 1000 mg/m^2 | Ixabepilone, 32 mg/m^2 + Capecitabine, 1000 mg/m^2 | Docetaxel, 75 mg/m^2 + Capecitabine, 1000 mg/m^2
Number analyzed (Participants) | 20 | 22 | 20
Participants
  Complete response (CR) | 1 | 1 | 0
  Partial response (PR) | 6 | 8 | 6
  Stable disease (SD) | 6 | 3 | 3
  Progressive disease (PD) | 4 | 9 | 9
  Discontinued before first tumor assessment | 3 | 0 | 1
  No tumor assessment due to other reasons | 0 | 0 | 1
  Unable to determine | 0 | 1 | 0

2. Secondary Outcome: Percentage of Triple-negative (TN) Participants With Best Response to Treatment of Complete or Partial
Description: The tumor response rate is defined as the total number of participants whose best response is CR or PR, divided by the number of randomized participants. Participants not evaluable for response are considered to be nonresponders. TN participants are those with tumors that do not express estrogen or progesterone receptors and that do not over express human epidermal growth factor receptor 2 (HER2).
Time Frame: Baseline to 6 weeks (end of Cycle 2)
Population: All TN participants who received ixabepilone plus capecitabine or docetaxel plus capecitabine.
Measure: Number; unit: Percentage of TN Participants
Arm/Group | Ixabepilone, 40 mg/m^2 + Capecitabine, 1000 mg/m^2 | Ixabepilone, 32 mg/m^2 + Capecitabine, 1000 mg/m^2 | Docetaxel, 75 mg/m^2 + Capecitabine, 1000 mg/m^2
Number analyzed (Participants) | 8 | 9 | 8
Percentage of TN Participants | 38 | 22 | 13

3. Secondary Outcome: Percentage of Nontriple-negative (NTN) Participants With Best Response to Treatment of Complete or Partial Per Cohort
Description: The tumor response rate is defined as the total number of participants whose best response is CR or PR, divided by the number of randomized participants. Participants not evaluable for response are considered to be nonresponders. NTN participants are who are not TN participants (TN participants are those with tumors that do not express estrogen or progesterone receptors and that do not overexpress HER2) and who received ixabepilone plus capecitabine or docetaxel plus capecitabine.
Time Frame: Baseline to 6 weeks (end of Cycle 2)
Population: All NTN participants who received ixabepilone plus capecitabine or docetaxel plus capecitabine.
Measure: Number; unit: Percentage of NTN Participants
Arm/Group | Ixabepilone, 40 mg/m^2 + Capecitabine, 1000 mg/m^2 | Ixabepilone, 32 mg/m^2 + Capecitabine, 1000 mg/m^2 | Docetaxel, 75 mg/m^2 + Capecitabine, 1000 mg/m^2
Number analyzed (Participants) | 12 | 13 | 12
Percentage of NTN Participants | 33 | 54 | 42

4. Secondary Outcome: Number of Participants With Death, Adverse Events (AEs), Drug-related AEs, Serious AEs (SAEs), Drug-related SAEs, AEs Leading to Discontinuation (AEDs), Drug-related AEDs, and Drug-related Peripheral Neuropathy
Description: An AE is any new untoward medical occurrence or worsening of a preexisting medical condition that does not necessarily have a causal relationship with this treatment. An SAE is any untoward medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency or abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Drug-related=possibly, probably, or certainly related or of unknown relationship to study treatment. Grade 3=Severe, Grade 4=Life-threatening.
Time Frame: Baseline to end of Cycle 1 (21 days), continuously
Population: All participants who received at least 1 dose of ixabepilone plus capecitabine or of docetaxel plus capecitabine.
Measure: Number; unit: Participants
Arm/Group | Ixabepilone, 40 mg/m^2 + Capecitabine, 1000 mg/m^2 | Ixabepilone, 32 mg/m^2 + Capecitabine, 1000 mg/m^2 | Docetaxel, 75 mg/m^2 + Capecitabine, 1000 mg/m^2
Number analyzed (Participants) | 20 | 22 | 20
Participants
  Deaths | 2 | 1 | 2
  AEs | 20 | 22 | 20
  Drug-related AEs | 20 | 22 | 19
  Drug-related AEs (Grade 3) | 8 | 9 | 8
  Drug-related AEs (Grade 4) | 6 | 3 | 6
  SAEs | 7 | 5 | 5
  Drug-related SAEs | 3 | 3 | 3
  Drug-related SAEs (Grade 3) | 2 | 2 | 2
  Drug-related SAEs (Grade 4) | 1 | 1 | 1
  AEDs | 4 | 9 | 4
  Drug-related AEDs | 2 | 7 | 3
  Drug-related AEDs (Grade 3) | 1 | 3 | 2
  Drug-related AEDs (Grade 4) | 1 | 1 | 0
  Drug-related peripheral neuropathy | 10 | 15 | 5
  Drug-related peripheral neuropathy (Grade 3) | 4 | 2 | 0
  Drug-related peripheral neuropathy (Grade 4) | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Abnormalities in Hematology Laboratory Results by Worst Common Terminology Criteria (CTC) Grade
Description: CTC Grade 1=Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2=Moderate; minimal, local or noninvasive intervention indicated. Grade 3=Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling. Grade 4=Life-threatening consequences; urgent intervention indicated.
Time Frame: Baseline in Cycle 1 (21 days) and then prior to start of each 21-day cycle
Population: All participants who received at least 1 dose of ixabepilone plus capecitabine or of docetaxel plus capecitabine.
Measure: Number; unit: Participants
Arm/Group | Ixabepilone, 40 mg/m^2 + Capecitabine, 1000 mg/m^2 | Ixabepilone, 32 mg/m^2 + Capecitabine, 1000 mg/m^2 | Docetaxel, 75 mg/m^2 + Capecitabine, 1000 mg/m^2
Number analyzed (Participants) | 20 | 22 | 20
Participants
  Neutropenia (Grades 1-4) | 18 | 15 | 17
  Neutropenia (Grade 3 or 4) | 12 | 10 | 15
  Leukopenia (Grades 1-4) | 20 | 19 | 17
  Leukopenia (Grade 3 or 4) | 9 | 9 | 12
  Thrombocytopenia (Grades 1-4) | 9 | 11 | 7
  Thrombocytopenia (Grade 3 or 4) | 0 | 1 | 0
  Anemia (Grades 1-4) | 18 | 21 | 17
  Anemia (Grade 3 or 4) | 0 | 1 | 0

6. Secondary Outcome: Number of Participants With Abnormalities in Serum Chemistry Laboratory Results
Description: ULN=Upper limit of normal among all laboratory ranges. Alanine aminotransferase (ALT) Grade 1:>ULN to 2.5*ULN; Grade 2: >2.5 to 5.0*ULN; Grade 3: >5.0 to 20.0*ULN; Grade 4: >20.0*ULN. Aspartate aminotransferase (AST) Grade 1: >ULN to 2.5*ULN; Grade 2: >2.5 to 5.0*ULN; Grade 3: >5.0 to 20.0*ULN; Grade 4: >20.0*ULN. Total bilirubin Grade 1: >ULN to 1.5*ULN; Grade 2: >1.5 to 3.0*ULN; Grade 3: >3.0 to 10.0*ULN; Grade 4: >10.0*ULN. Creatine Grade 1: >ULN to 1.5*ULN; Grade 2: 1.5 to 3.0*ULN; Grade 3: >3.0 to 6.0*ULN; Grade 4: >6.0*ULN.
Time Frame: Baseline in Cycle 1 (21 days) and then prior to start of each 21-day cycle
Population: All participants who received at least 1 dose of ixabepilone plus capecitabine or of docetaxel plus capecitabine.
Measure: Number; unit: Participants
Arm/Group | Ixabepilone, 40 mg/m^2 + Capecitabine, 1000 mg/m^2 | Ixabepilone, 32 mg/m^2 + Capecitabine, 1000 mg/m^2 | Docetaxel, 75 mg/m^2 + Capecitabine, 1000 mg/m^2
Number analyzed (Participants) | 20 | 22 | 20
Participants
  ALT, high (Grades 1-4) | 4 | 3 | 5
  ALT, high (Grade 3 or 4) | 0 | 0 | 0
  AST, high (Grades 1-4) | 7 | 5 | 5
  AST, high (Grade 3 or 4) | 0 | 0 | 0
  Total bilirubin, high (Grades 1-4) | 0 | 1 | 0
  Total bilirubin, high (Grade 3 or 4) | 0 | 0 | 0
  Creatinine, high (Grades 1-4) | 1 | 1 | 2
  Creatinine, high (Grade 3 or 4) | 0 | 0 | 0

7. Secondary Outcome: Time to Progression
Description: Time to progression is defined as the time from date of randomization until the date that PD is first reported. Participants who die without a reported prior progression are considered to have progressed on the day of their death. Those who did not progress or die are censored at the day of their last tumor assessment.
Time Frame: Baseline to date progressive disease reported
Population: This study was terminated due to inadequate enrollment. Consequently, time to progression was not analyzed.
Arm/Group | Ixabepilone, 40 mg/m^2 + Capecitabine, 1000 mg/m^2 | Ixabepilone, 32 mg/m^2 + Capecitabine, 1000 mg/m^2 | Docetaxel, 75 mg/m^2 + Capecitabine, 1000 mg/m^2
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Duration of Response
Description: Duration of overall response is computed for participants whose best response is either PR or CR and is measured from the time measurement criteria are first met for CR or PR (whichever status is recorded first) until the first date of documented PD or death. Participants who did not relapse or die are censored on the date of their last tumor assessment.
Time Frame: Baseline (date of randomization) to date CR or PR criteria first met
Population: This study was terminated due to inadequate enrollment. Consequently, duration of response was not analyzed.
Arm/Group | Ixabepilone, 40 mg/m^2 + Capecitabine, 1000 mg/m^2 | Ixabepilone, 32 mg/m^2 + Capecitabine, 1000 mg/m^2 | Docetaxel, 75 mg/m^2 + Capecitabine, 1000 mg/m^2
Number analyzed (Participants) | 0 | 0 | 0

9. Primary Outcome: Percentage of Participants With Best Response to Treatment of Complete or Partial
Description: The tumor response rate is defined as the number of participants with a best tumor response of CR or PR (as assessed by the investigator according to RECIST criteria), divided by the number of participants randomized in that arm.
Time Frame: Baseline to 6 weeks (end of Cycle 2)
Population: All participants with measurable disease who have a correct cancer diagnosis and have received any treatment.
Measure: Number; unit: Percentage of patients
Arm/Group | Ixabepilone, 40 mg/m^2 + Capecitabine, 1000 mg/m^2 | Ixabepilone, 32 mg/m^2 + Capecitabine, 1000 mg/m^2 | Docetaxel, 75 mg/m^2 + Capecitabine, 1000 mg/m^2
Number analyzed (Participants) | 20 | 22 | 20
Percentage of patients | 35 | 41 | 30

10. Secondary Outcome: Median Number of Treatment Cycles
Description: The first dosing date is defined as the date of the first dose of chemotherapy or capecitabine, whichever was administered first. Cycles are defined as the time from Day 1 of the cycle until the day before the next cycle. The last cycle per participant is the 21-day period following Day 1 of that cycle.
Time Frame: Day 1 to end of Cycle 18, maximum (54 weeks)
Population: All participants who received at least 1 dose of ixabepilone plus capecitabine or of docetaxel plus capecitabine.
Measure: Median (Full Range); unit: Treatment cycles
Arm/Group | Ixabepilone, 40 mg/m^2 + Capecitabine, 1000 mg/m^2 | Ixabepilone, 32 mg/m^2 + Capecitabine, 1000 mg/m^2 | Docetaxel, 75 mg/m^2 + Capecitabine, 1000 mg/m^2
Number analyzed (Participants) | 20 | 22 | 20
Treatment cycles | 3.0 [1 to 16] | 4.5 [1 to 18] | 6.0 [1 to 17]

ADVERSE EVENTS:
Arm/Group | Docetaxel | Ixabepilone 32 | Ixabepilone 40
Serious Adverse Events (participants affected / at risk) | 5/20 | 5/22 | 7/20
Other Adverse Events (participants affected / at risk) | 20/20 | 22/22 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel (N=20) | Ixabepilone 32 (N=22) | Ixabepilone 40 (N=20)
BLOOD CREATININE INCREASED (Investigations) | 0 | 0 | 1
NEUTROPHIL COUNT DECREASED (Investigations) | 0 | 0 | 1
EMBOLISM (Vascular disorders) | 0 | 0 | 1
HYPOTENSION (Vascular disorders) | 1 | 0 | 0
HEADACHE (Nervous system disorders) | 0 | 0 | 1
DIZZINESS (Nervous system disorders) | 0 | 1 | 0
SOMNOLENCE (Nervous system disorders) | 0 | 1 | 0
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 0 | 1 | 0
NAUSEA (Gastrointestinal disorders) | 0 | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 0 | 2 | 1
COLONIC OBSTRUCTION (Gastrointestinal disorders) | 0 | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 1 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 1 | 2
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0
ELECTROLYTE IMBALANCE (Metabolism and nutrition disorders) | 0 | 1 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 1 | 0
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 2 | 0 | 0
INCISION SITE PAIN (Injury, poisoning and procedural complications) | 0 | 1 | 0
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
ASTHENIA (General disorders) | 0 | 1 | 0
OEDEMA PERIPHERAL (General disorders) | 0 | 1 | 0
CATHETER THROMBOSIS (General disorders) | 0 | 0 | 1
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel (N=20) | Ixabepilone 32 (N=22) | Ixabepilone 40 (N=20)
DRY EYE (Eye disorders) | 0 | 0 | 1
PHOTOPHOBIA (Eye disorders) | 1 | 0 | 0
VISION BLURRED (Eye disorders) | 0 | 2 | 0
VISUAL IMPAIRMENT (Eye disorders) | 1 | 0 | 0
LACRIMATION INCREASED (Eye disorders) | 3 | 1 | 1
OCULAR SURFACE DISEASE (Eye disorders) | 0 | 0 | 1
WEIGHT DECREASED (Investigations) | 3 | 2 | 5
HAEMOGLOBIN DECREASED (Investigations) | 2 | 10 | 5
BLOOD GLUCOSE INCREASED (Investigations) | 0 | 2 | 0
PLATELET COUNT DECREASED (Investigations) | 0 | 3 | 1
BLOOD CREATININE INCREASED (Investigations) | 0 | 0 | 1
EOSINOPHIL COUNT DECREASED (Investigations) | 1 | 0 | 0
NEUTROPHIL COUNT DECREASED (Investigations) | 3 | 2 | 5
EJECTION FRACTION DECREASED (Investigations) | 1 | 0 | 0
GRANULOCYTE COUNT DECREASED (Investigations) | 1 | 0 | 1
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 3 | 5 | 4
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 1 | 0 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 1 | 2
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 2 | 3
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 | 3 | 0
TACHYCARDIA (Cardiac disorders) | 1 | 0 | 0
PALPITATIONS (Cardiac disorders) | 1 | 0 | 0
SINUS TACHYCARDIA (Cardiac disorders) | 0 | 0 | 2
FLUSHING (Vascular disorders) | 0 | 0 | 1
HOT FLUSH (Vascular disorders) | 0 | 3 | 0
HYPOTENSION (Vascular disorders) | 1 | 1 | 0
LYMPHOEDEMA (Vascular disorders) | 1 | 1 | 1
HYPERTENSION (Vascular disorders) | 1 | 0 | 1
VENOUS THROMBOSIS (Vascular disorders) | 1 | 0 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 | 0 | 0
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 0 | 0 | 1
ANXIETY (Psychiatric disorders) | 3 | 3 | 1
INSOMNIA (Psychiatric disorders) | 1 | 4 | 0
DEPRESSION (Psychiatric disorders) | 1 | 3 | 2
HYPERSENSITIVITY (Immune system disorders) | 2 | 0 | 0
HEADACHE (Nervous system disorders) | 4 | 3 | 3
MIGRAINE (Nervous system disorders) | 1 | 0 | 0
DIZZINESS (Nervous system disorders) | 1 | 1 | 3
DYSGEUSIA (Nervous system disorders) | 2 | 3 | 3
PARAESTHESIA (Nervous system disorders) | 0 | 2 | 1
HYPOAESTHESIA (Nervous system disorders) | 1 | 2 | 0
COGNITIVE DISORDER (Nervous system disorders) | 0 | 0 | 1
NEUROPATHY PERIPHERAL (Nervous system disorders) | 3 | 7 | 2
EXTRAPYRAMIDAL DISORDER (Nervous system disorders) | 0 | 0 | 1
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 3 | 8 | 7
NAUSEA (Gastrointestinal disorders) | 10 | 17 | 8
VOMITING (Gastrointestinal disorders) | 4 | 8 | 6
DIARRHOEA (Gastrointestinal disorders) | 8 | 12 | 9
DYSPEPSIA (Gastrointestinal disorders) | 2 | 5 | 1
DYSPHAGIA (Gastrointestinal disorders) | 2 | 2 | 0
GASTRITIS (Gastrointestinal disorders) | 1 | 0 | 0
FLATULENCE (Gastrointestinal disorders) | 1 | 0 | 1
STOMATITIS (Gastrointestinal disorders) | 4 | 4 | 5
CONSTIPATION (Gastrointestinal disorders) | 5 | 7 | 12
HAEMORRHOIDS (Gastrointestinal disorders) | 0 | 0 | 1
LIP SWELLING (Gastrointestinal disorders) | 0 | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 3 | 1
FAECAL INCONTINENCE (Gastrointestinal disorders) | 1 | 0 | 0
NEUTROPENIC COLITIS (Gastrointestinal disorders) | 0 | 0 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 2 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 | 0 | 0
EAR PAIN (Ear and labyrinth disorders) | 0 | 0 | 1
INFECTION (Infections and infestations) | 0 | 0 | 1
PNEUMONIA (Infections and infestations) | 0 | 0 | 1
SINUSITIS (Infections and infestations) | 1 | 1 | 2
BRONCHITIS (Infections and infestations) | 0 | 1 | 1
CANDIDIASIS (Infections and infestations) | 1 | 0 | 0
NAIL INFECTION (Infections and infestations) | 1 | 1 | 1
ORAL CANDIDIASIS (Infections and infestations) | 1 | 0 | 0
LOCALISED INFECTION (Infections and infestations) | 1 | 0 | 0
FUNGAL SKIN INFECTION (Infections and infestations) | 0 | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 1 | 1 | 0
NAIL BED INFECTION FUNGAL (Infections and infestations) | 1 | 0 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 2
POLLAKIURIA (Renal and urinary disorders) | 0 | 1 | 1
BLADDER SPASM (Renal and urinary disorders) | 0 | 0 | 1
STRESS URINARY INCONTINENCE (Renal and urinary disorders) | 1 | 0 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 4 | 2
HYPOKALAEMIA (Metabolism and nutrition disorders) | 2 | 6 | 4
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 | 1 | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 2 | 2
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 2 | 1 | 3
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 1 | 2 | 1
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 6 | 7 | 6
ANAEMIA (Blood and lymphatic system disorders) | 4 | 6 | 2
LEUKOPENIA (Blood and lymphatic system disorders) | 6 | 2 | 3
LYMPHOPENIA (Blood and lymphatic system disorders) | 3 | 0 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 11 | 5 | 5
MONOCYTOPENIA (Blood and lymphatic system disorders) | 1 | 0 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 | 0 | 0
RASH (Skin and subcutaneous tissue disorders) | 2 | 4 | 2
ALOPECIA (Skin and subcutaneous tissue disorders) | 4 | 10 | 6
DRY SKIN (Skin and subcutaneous tissue disorders) | 2 | 1 | 2
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 1 | 2 | 2
KOILONYCHIA (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
ONYCHOLYSIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
ONYCHOCLASIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 4 | 2 | 3
ONYCHOMADESIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
PALMAR ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
EXFOLIATIVE RASH (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
SKIN EXFOLIATION (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
SKIN DISCOLOURATION (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 8 | 12 | 8
BREAST DISCHARGE (Reproductive system and breast disorders) | 0 | 0 | 1
PELVIC HAEMATOMA (Reproductive system and breast disorders) | 0 | 0 | 1
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 | 0 | 1
MENSTRUATION IRREGULAR (Reproductive system and breast disorders) | 0 | 1 | 1
LIMB INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0
WOUND SECRETION (Injury, poisoning and procedural complications) | 0 | 0 | 1
WOUND COMPLICATION (Injury, poisoning and procedural complications) | 0 | 0 | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1
BONE PAIN (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 | 3 | 1
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
JOINT STIFFNESS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3 | 1 | 5
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 | 3 | 3
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 2
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 4
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
PAIN (General disorders) | 3 | 2 | 1
CHILLS (General disorders) | 1 | 2 | 0
OEDEMA (General disorders) | 1 | 0 | 1
FATIGUE (General disorders) | 12 | 17 | 15
PYREXIA (General disorders) | 5 | 1 | 3
XEROSIS (General disorders) | 1 | 0 | 0
ASTHENIA (General disorders) | 1 | 0 | 0
FIBROSIS (General disorders) | 0 | 0 | 1
CHEST PAIN (General disorders) | 1 | 1 | 1
OEDEMA PERIPHERAL (General disorders) | 2 | 5 | 4
CATHETER SITE PAIN (General disorders) | 1 | 0 | 0
CATHETER THROMBOSIS (General disorders) | 0 | 0 | 1
MUCOSAL INFLAMMATION (General disorders) | 6 | 3 | 3
CATHETER SITE ERYTHEMA (General disorders) | 1 | 0 | 0
INFLUENZA LIKE ILLNESS (General disorders) | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.